CLINICAL TRIAL: NCT06602596
Title: Hoosier Sport: Refining and Implementing a Sustainable Campus-Community Partnership in Rural Indiana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Kyle A. Kercher, Assistant Professor, Indiana University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 23985
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: CVD; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group in the Hoosier Sport study consists of students who are not enrolled in the PE class and therefore do not participate in the Hoosier Sport program. These students continue with their regular school activities without the added sport, leadership, and health education components provided in the intervention.
- Test group - Hoosier Sport Participants (Experimental): The intervention group in the Hoosier Sport study consists of students enrolled in the PE class who actively participate in the Hoosier Sport program. These students engage in an 8-week curriculum that includes unique sports activities, leadership exercises, and health education sessions designed to promote physical activity and well-being.
  Interventions: Behavioral: Hoosier Sport

INTERVENTIONS:
Behavioral: Hoosier Sport — The Hoosier Sport intervention is an 8-week program designed for students in PE classes, focusing on enhancing physical activity and promoting health through sport. The curriculum includes unique sports activities, leadership exercises, and health education, aimed at improving students' physical and psychological well-being. The program also addresses the effects of screen time and social media on physical activity, encouraging healthier behaviors. Throughout the intervention, students wear AX3 accelerometers to track changes in their physical activity levels, helping to assess the program's impact.
  Arms: Test group - Hoosier Sport Participants

SUMMARY:
Hoosier Sport is a sport-based youth development program that uses the power of sport to teach children and adolescents sport and leadership skills while promoting health education. Conducted in rural middle and high schools, the program aims to enhance health and wellness by incorporating unique sports such as volleyball and flag football, along with leadership activities like goal setting and health education on the importance of exercise and a healthy lifestyle. The program runs for eight weeks each semester (Fall and Spring), with sessions twice a week during PE class, where college service-learning students lead the curriculum. Data on physical activity and psychosocial factors are collected to assess changes in health, ensuring confidentiality through strict IRB protocols.

DETAILED DESCRIPTION:
Hoosier Sport is a comprehensive sport-based youth development program designed to enhance the health and wellness of rural children and adolescents. The program leverages the power of sport to teach essential sport skills, leadership qualities, and promote health education. Conducted primarily in physical education (PE) classes, with occasional sessions in health classes, Hoosier Sport spans eight weeks with sessions twice a week. The curriculum focuses on unique sports such as strength training, pickleball, and flag football, and integrates activities that foster leadership (e.g., goal setting) and health education (e.g., the importance of regular exercise and a healthy lifestyle).

A key objective of Hoosier Sport is to explore how participation in sports can satisfy the basic psychological needs of autonomy, competence, and relatedness. By providing structured yet flexible activities that allow for individual achievement and peer interaction, the program aims to enhance students' intrinsic motivation to engage in physical activity. Additionally, Hoosier Sport addresses the growing concern of screen time and social media usage, which are known to negatively impact physical activity levels. The program integrates discussions and activities that encourage students to reflect on their screen time habits, understand the effects of social media on body image and activity levels, and develop healthier behaviors.

To objectively measure the impact of the program on physical activity (PA), Hoosier Sport utilizes advanced accelerometers (AX3 devices). These devices are worn by students for a week at a time, capturing detailed data on their physical activity patterns. This data allows the research team to accurately assess changes in PA levels throughout the program, providing insights into the effectiveness of the intervention. Alongside physical activity, the program collects data on psychosocial factors, such as self-esteem and social skills, to identify broader health and behavioral outcomes. Exploratory data includes screen time, social media usage, as well as inhibitory control. All collected data is handled anonymously, following strict Institutional Review Board (IRB) protocols to ensure the privacy and protection of participants. Through this multifaceted approach, Hoosier Sport aims not only to improve physical health but also to foster psychological well-being and sustainable healthy behaviors among rural youth.

ELIGIBILITY:
Inclusion Criteria:

* Must provide parental consent and student assent.
* Enrollment in a physical education class

Exclusion Criteria:

-Presence of medical conditions or physical limitations that prevent safe participation in physical activity, as determined by the Physical Activity Readiness Questionnaire (PAR-Q) or a medical professional.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-05-08 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
Feasibility of Intervention Measure (FIM) | Measured at week 0 and week 9
  How feasible the intervention was from the perspective of the participants. This is measured through questionnaire.
Acceptability of Intervention Measure (IAM) | Measured at week 0 and week 9
  How acceptable the intervention is to the participants. This is measured through questionnaire.
Intervention Appropriateness Measure (AIM) | Measured at week 0 and week 9
  How appropriate the intervention is to the participants. This is measured through questionnaire.

SECONDARY OUTCOMES:
Daily Total Physical Activity of Participants | Week 1 (for 7 days), and week 9 (for 7 days)
  Accelerometers (Axivity - AX3 model) will be used to track daily total physical activity
Heart Rate of Participants | HR will be taken at week 0 and week 9 before and following the 6-minute walk test.
  heart rate measured via a blood pressure monitor
Blood Pressure of Participants | BP will be taken at week 0 and week 9 before and following the 6-minute walk test.
  Blood pressure measured via a blood pressure monitor
Basic Psychological Needs of Participants in Intervention Environment | Assessed at week 0 and week 9
  Basic Psychological Needs and Satisfaction and Frustration scale (BPNSF). This entails feelings/perceptions of autonomy, relatedness, competence, enjoyment, satisfaction, and frustration in the study setting.
Physical Literacy of Participants | Assessed at week 0 and week 9
  the Canadian Assessment of Physical Literacy second addition (CAPL-2) will be used. A higher score on the CAPL-2 indicates higher physical literacy.
Cardiovascular Fitness Levels of Participants | Assessed at week 0 and week 9
  the 6-minute walk test will be used to assess changes in fitness. Greater distance walked in the 6 minute time frame is related to greater levels of cardiovascular fitness.
Muscular Endurance Levels of Participants | Assessed at week 0 and week 9
  The plank test will be used to assess changes in fitness. The longer the plank is held, the greater the muscular endurance of the participant.
Policy, Systems, and Environmental Factors Influencing Participant Physical Activity and Nutrition Behavior. | Assessed at week 0 and week 9
  a survey will collect data on Policy, Systems and Environmental (PSE) changes using a 5 questions guided by the SNAP-Ed curriculum. Higher scores will indicate better PSE support for physical activity and healthy nutrition opportunities for the participants in their school environment.

OTHER OUTCOMES:
Daily screen time | Assessed at week 0 and week 9
  data from participants' phone settings will be used to capture daily screen time. Participants will navigate to their screen time settings, where a comprehensive and objective report of their weekly screen time (including average daily screen time) is available. Here, participants will screenshot this data and airdrop it to a secured IU dropbox location.
Daily social media usage | Assessed at week 0 and week 9
  data from participants' phone settings will be used to capture daily screen time. Participants will navigate to their screen time settings, where a comprehensive and objective report of their weekly screen time (including average daily social media usage) is available. Here, participants will screenshot this data and airdrop it to a secured IU dropbox location.
Social media addiction | Assessed at week 0 and week 9
  participants will complete the Bergen Social Media Addiction Scale to assess social media addiction.
Inhibitory control | Assessed at week 0 and week 9
  The Color-Word trial from the Stroop Color and Word Test will be delivered on an iPad/tablet to participants to measure inhibitory control.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Indiana University, Bloomington, Indiana
  - White River Valley Middle School, Lyons, Indiana

IPD SHARING:
Plan to Share IPD: No